CLINICAL TRIAL: NCT05836831
Title: Indian Trial of Tranexamic Acid in Spontaneous Intracerebral Haemorrhage
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Christian Medical College and Hospital, Ludhiana, India (Other)
Collaborators: Indian Council of Medical Research (Other Government); Sree Chitra Tirunal Institute for Medical Sciences & Technology (Other Government); Post Graduate Institute of Medical Education and Research, Chandigarh (Other); St. Stephen's Hospital, Delhi (Other); All India Institute of Medical Sciences (Other); Amrita Institute of Medical Sciences & Research Center (Other); Kasturba Medical College Manipal, India (Unknown); Institute of Neurosciences Kolkata (Other); Bangur Institute of Neurosciences Kolkata, India (Unknown); Guwahati Neurological Research Center, Guwahati, India (Unknown); Baptist Christian Hospital, Tezpur, India (Unknown); National Institute of Mental Health and Neuro Sciences, India (Other); Jawaharlal Institute of Postgraduate Medical Education & Research (Other Government); Christian Medical College, Vellore, India (Other); CARE Hospitals Hyderabad, India (Unknown); Lalitha Super Specialities Hospital Guntur, India (Unknown); Dr. Ramesh Cardiac and Multispeciality Hospital Guntur, India (Unknown); Government General Hospital Guntur, India (Unknown); Fortis Escorts Hospital Jaipur, India (Unknown); Institute of Medical Sciences of the Banaras Hindu University, India (Other); Atal Institute of Medical Super Specilities, (AIMSS) Chamiana, Shimla (Unknown); All India Institute of Medical Sciences, Bhubaneswar (Other); KLEs Dr. Prabhakar Kore Hospital & Medical Research Centre Balgaum, India (Unknown); Guru Gobind Singh Medical College & Hospital (Other); PBM Hospital Bikaner, India (Unknown); Shree Krishna Hospital Pramukhswami Medical College Anand, India (Unknown); Apollo Excelcare Hospitals Guwahati, India (Unknown); Manipal Hospital Bangalore, India (Unknown); Artemis Hospital Gurgaon, India (Unknown); Dr. Kamakshi Memorial Hospital Chennai, India (Unknown); Bharati Vidyapeeth DTU Medical College Pune, India (Unknown); Aster MIMS Hospital Calicut, India (Unknown); Holy Spirit Hospital Mumbai, India (Unknown); Sparsh Superspeciality Hospital Bangalore, India (Unknown); King George's Medical University, Lucknow, India (Unknown); Assam Medical College, Dibrugarh, India (Unknown); KG Hospital and Post Graduate Medical Institute Coimbatore, India (Unknown); Tirunelveli Medical College, Tirunelveli, India (Unknown); Santokba Durlabhji Memorial Hospital, Jaipur, India (Unknown); Tezpur Medical College and Hospital, Assam, India (Unknown); Baby Memorial Hospital Calicut, India (Unknown); Institute of Human Behaviour and Allied Sciences Delhi, India (Unknown); The Calcutta Medical Research Institute, Kolkata, India (Unknown); Fortis Hospital Mulund Mumbai, India (Unknown); Government Medical College Trivandrum, India (Unknown); Ruby Hall Clinic, Pune, India (Unknown); Manipal Hospital Goa, India (Unknown)
Responsible Party: Principal Investigator, Jeyaraj D Pandian, Principal and Professor, Department of Neurology, Christian Medical College and Hospital, Ludhiana, India
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: INTRINSIC Trial
Record Dates: First submitted 2023-04-19; First posted 2023-05-01 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Intracerebral Hemorrhagic Stroke
Keywords: Stroke; Spontaneous Intracerebral Haemorrhage; Tranexamic acid
MeSH Terms: conditions — Hemorrhagic Stroke; Stroke | interventions — Tranexamic Acid

STUDY DESIGN:
Intervention Model Description: Multicentric, randomized, open-label, clinical trial
Who Masked: Participant
Masking Description: Open-label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): The treatment arm will consist of giving intravenously 2 grams of Tranexamic Acid in 100 ml sodium chloride 0.9 % administered over 45 minutes. Intensive systolic blood pressure reduction to less than 140 mmHg will be done using antihypertensive agents (intravenous and/or oral) which is to be achieved within one hour and has to be maintained over seven days. BP monitoring is done every 15 minutes in the first hour and thereafter every hour for the next six hours after the initiation of intensive BP control. The choice of antihypertensive will depend on the clinician's preference.
  Interventions: Drug: Tranexamic acid injection
- Control Arm (No Intervention): The control arm will receive a standard of care management as per the institutional practice. Intensive systolic blood pressure reduction to less than 140 mmHg will be done using antihypertensive (intravenous and/or oral) which is to be achieved within one hour and has to be maintained over seven days. BP monitoring is done for every 15 minutes in the first hour and thereafter every hour for the next six hours after the initiation of intensive BP control. The choice of antihypertensive will depend on the clinician's preference.

INTERVENTIONS:
Drug: Tranexamic acid injection — The treatment arm will consist of giving intravenously 2 grams of Tranexamic Acid in 100 ml sodium chloride 0.9 % administered over 45 minutes.
  Other Names: Injection Pause 500 mg/5 ml; Injection Cyklokapron 500 mg/5 ml; Injection Trapic 500 mg/5 ml; Injection Tramix 500 mg/5 ml
  Arms: Intervention Arm

SUMMARY:
This multicenter, pragmatic randomized, open-label clinical trial aims to assess whether Tranexamic Acid improves outcomes in adult patients with spontaneous intracerebral haemorrhage.

The participants presenting within 4.5 hours of the onset of symptoms of stroke with intracerebral haemorrhage confirmed on Computed Tomography (CT Scan) will be randomized into two groups in a 1:1 ratio using a central online randomization. The treatment arm will consist of giving intravenously 2 grams of Tranexamic Acid in 100 ml 0.9% sodium chloride administered over 45 minutes. Control arm patients will receive standard of care treatment as per the institutional protocol. In both arms, intensive systolic blood pressure reduction to less than 140 mmHg will be done using antihypertensive medications, which has to be achieved within one hour and will be maintained over next seven days. The choice of antihypertensive drug will depend on the clinician's preference.

Both groups will have a repeat CT scan after 24 hours to check for any increase in the haematoma volume. Any deterioration in the neurological status will warrant urgent brain imaging. On day 7, the patient will be assessed for their NIHSS score and mRS score. On day 90, quality of life and the functional outcome will be assessed.

DETAILED DESCRIPTION:
Global Burden of Disease, Injury and Risk factors for hemorrhagic stroke 2010 estimated the burden of spontaneous intracranial haemorrhage (sICH) in India is profound (32 -49%) and it is associated with high mortality (up to 63 %) due to haematoma expansion which occurs in 38% of ICH within first few hours of presentation. Early administration of haemostatic drugs has been used in patients with trauma and was associated with improved outcomes. Similarly, if haemostatic drugs are administered early, which can be a simple and cost-effective intervention, may improve the functional outcomes in patients with sICH. Recently, the Tranexamic acid for hyperacute primary IntraCerebral Haemorrhage (TICH 2 trial), which was done to see the effectiveness of the administration of tranexamic acid on hematoma expansion and functional outcomes at three months in patients who presented with sICH within 8 hours of presentation of symptoms onset, showed a decrease in haematoma expansion but no improvement in functional outcome at 90 days. Further larger randomized control trials are required to ascertain the effect of early administration of Tranexamic acid (TXA) in sICH. In India patients present to hospitals in the early stages that have developed symptoms after sICH and we propose to study the effect of intravenous Tranexamic Acid for hyperacute primary intracerebral haemorrhage within 4.5 hours of sICH.

Trial Population:

This multi-centric study will be conducted at 50 stroke centres in India associated with the INSTRuCT Network. All patients presenting with symptoms of stroke to the hospital and admitted to the stroke units will be screened for eligibility and if met, will be included in the study. The INTRINSIC trial intends to recruit 3400 patients.

Trial Design:

INTRINSIC Trial will be a multicenter, randomized, open-label, clinical trial. The participants will be randomized into two groups in a 1:1 ratio using a central database of INSTRuCT central online randomization. The baseline characteristics will be adjusted to stroke severity using the NIHSS score and the volume of haematoma. The treatment arm will consist of giving intravenously 2 grams of Tranexamic Acid in 100 ml sodium chloride 0.9 % administered over 45 minutes. Control arm patients will receive standard of care management as per the institutional protocol. Both groups will have a repeat CT scan after 24 hours to check for any increase in the haematoma volume. Any deterioration in the Glasgow Coma Scale (GCS) will warrant urgent brain CT scans. Antihypertensive drugs used and their doses to control BP will be recorded for up to 7 days. On day 7, the patient will be assessed for their NIHSS score and mRS score. On day 90, quality of life and the functional outcome will be assessed.

The need for this study:

The proportion of ICH is high in India and other LMIC's, particularly in Asia. Currently, there are no effective treatments available for sICH. Moreover, Tranexamic Acid is cheap, easily available and easy to administer.

ELIGIBILITY:
Inclusion Criteria:

Adult patients aged more than 18 years, presenting with non- traumatic intracerebral haemorrhage within 4.5 hours of onset of stroke symptoms

Exclusion Criteria:

1. Patients with ICH secondary to anticoagulation, thrombolysis, or known underlying structural abnormality such as arteriovenous malformation, aneurysm, tumor, venous thrombosis or due to known hereditary coagulation disorders.
2. Contraindication to TXA.
3. Concurrent participation in another trial.
4. Pre-stroke life expectancy <3 months (e.g. advanced metastatic cancer).
5. Glasgow coma scale (GCS) ⩽5.
6. ICH secondary to trauma.
7. Women of childbearing potential, pregnant, or breastfeeding at randomization.
8. Geographical or other factors that prohibit follow-upto 90 days.
9. Concurrent or planned treatment with any other hemostatic agents.
10. ICH volume >60 mL as measured by ABC/2 method.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3400 (Estimated)
Dates: Start 2022-08-30 (Actual); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Death | 30 days
  Death at day 30. Absolute difference of 3% between intervention and control arm for the number of participants that expired at day 30

SECONDARY OUTCOMES:
Change in hematoma volume | 24 hours
  Radiological (CT scan): Change in hematoma volume from baseline to 24 hours scan, hematoma location and new infraction
Neurological impairment | 7 days
  Neurological impairment National Institutes of Health Stroke Scale (NIHSS) at day 7 (or discharge if sooner). Lower NIHSS indicates a good outcome.
modified Rankin Scale (mRS) | 90 days
  Dependency using the seven-level modified Rankin Scale (mRS) at day 90. Good outcome is 0-2 and bad outcome is 3-6. Lower mRS indicated good outcome.
Quality of life EQ-5D | 90 days
  Quality of life EuroQoL-5 dimension (EQ-5D) at day 90. Lover score indicates good outcome

CONTACTS AND LOCATIONS:
Overall Officials: Jeyaraj D Pandian, MD DM, Principal Investigator — Christian Medical College and Hospital, Ludhiana, Punjab, India
Locations (48):
- India (48):
  - Government General Hospital, Guntur, Andhra Pradesh
  - Lalitha Super Specialty Hospital, Guntur, Andhra Pradesh
  - Dr Ramesh Cardiac and Multispecialty Hospital, Guntur, Andhra Pradesh
  - Assam Medical College, Dibrugarh, Assam
  - Guwahati Neurological Research Center, Guwahati, Assam
  - Apollo Excelcare Hospitals, Guwahati, Assam
  - Baptist Christian Hospital, Tezpur, Assam
  - Tezpur Medical College and Hospital, Tezpur, Assam
  - Manipal Hospital, Panjim, Goa
  - Shree Krishna Hospital Pramukhswami Medical College, Anand, Gujarat
  - Artemis Hospital, Gurgaon, Haryana
  - All India Institute of Medical Sciences, Bilāspur, Himachal Pradesh
  - Atal Institute of Medical Super Specilities, (AIMSS) Chamiana, Shimla, Himachal Pradesh
  - Manipal Hospital, Bangalore, Karnataka
  - Sparsh Superspeciality Hospital, Bangalore, Karnataka
  - National Institute of Mental Health and Neuro-Sciences, Bangalore, Karnataka
  - KLE's Dr. Prabhakar Kore Hospital & Medical Research Centre, Belagavi, Karnataka
  - Kasturba Medical College Manipal, Manipal, Karnataka
  - Baby Memorial Hospital, Calicut, Kerala
  - ASTER MIMS Hospital, Calicut, Kerala
  - Amrita Institute for Medical Sciences and Research Center, Kochi, Kerala
  - Government Medical College Trivandrum, Thiruvananthapuram, Kerala
  - Sree Chitra Tirunal Institute for Medical Sciences and Technology, Thiruvananthapuram, Kerala
  - Fortis Hospital Mulund, Mumbai, Maharashtra
  - Holy Spirit Hospital, Mumbai, Maharashtra
  - Ruby Hall Clinic, Pune, Maharashtra
  - Bharati Vidyapeeth DTU Medical College, Pune, Maharashtra
  - All India Institute of Medical Sciences, New Delhi, National Capital Territory of Delhi
  - Institute of Human Behaviour and Allied Sciences, New Delhi, National Capital Territory of Delhi
  - All India Institute of Medical Sciences, Bhubaneswar, Odisha
  - Guru Gobind Singh Medical College and Hospital, Farīdkot, Punjab
  - Christian Medical College and Hospital, Ludhiana, Punjab, Ludhiana, Punjab
  - PBM Hospital, Bikaner, Rajasthan
  - Santokba Durlabhji Memorial Hospital, Jaipur, Rajasthan
  - Fortis Escorts Hospital, Jaipur, Rajasthan
  - Dr. Kamakshi Memorial Hospital, Chennai, Tamil Nadu
  - KG Hospital and Post Graduate Medical Institute Coimbatore, Coimbatore, Tamil Nadu
  - Jawaharlal Institute of Postgraduate Medical Education and Research, Puducherry, Tamil Nadu
  - Tirunelveli Medical College, Tirunelveli, Tamil Nadu
  - Christian Medical College Vellore, Vellore, Tamil Nadu
  - CARE Hospitals, Hyderabad, Telangana
  - King George's Medical University, Lucknow, Uttar Pradesh
  - Institute of Medical Sciences of the Banaras Hindu University (BHU), Varanasi, Uttar Pradesh
  - Institute of Neurosciences, Kolkata, West Bengal
  - Bangur Institute of Neurosciences, Kolkata, West Bengal
  - The Calcutta Medical Research Center, Kolkata, West Bengal
  - Postgraduate Institute for Medical Education and Research, Chandigarh
  - St Stephen's Hospital, Delhi

IPD SHARING:
Plan to Share IPD: No
All information collected from medical records for the study will be stored electronically in a specifically designed database at the Christian Medical College and Hospital, Ludhiana, Punjab, India. Participants information will be identified only by their initials and a study registration number. Any information transferred electronically will be coded to protect confidentiality. All computer records will be password-protected. The study results may be presented at conferences or in scientific publications, but individual participants will not be identifiable. If needed, data will be available in future for other researchers outside the primary research group for secondary purposes, such as meta-analyses, reanalysis, or replication of results.

REFERENCES:
- [Background] Sprigg N, Flaherty K, Appleton JP, Al-Shahi Salman R, Bereczki D, Beridze M, Christensen H, Ciccone A, Collins R, Czlonkowska A, Dineen RA, Duley L, Egea-Guerrero JJ, England TJ, Krishnan K, Laska AC, Law ZK, Ozturk S, Pocock SJ, Roberts I, Robinson TG, Roffe C, Seiffge D, Scutt P, Thanabalan J, Werring D, Whynes D, Bath PM; TICH-2 Investigators. Tranexamic acid for hyperacute primary IntraCerebral Haemorrhage (TICH-2): an international randomised, placebo-controlled, phase 3 superiority trial. Lancet. 2018 May 26;391(10135):2107-2115. doi: 10.1016/S0140-6736(18)31033-X. Epub 2018 May 16. PMID 29778325
- [Background] Meretoja A, Churilov L, Campbell BC, Aviv RI, Yassi N, Barras C, Mitchell P, Yan B, Nandurkar H, Bladin C, Wijeratne T, Spratt NJ, Jannes J, Sturm J, Rupasinghe J, Zavala J, Lee A, Kleinig T, Markus R, Delcourt C, Mahant N, Parsons MW, Levi C, Anderson CS, Donnan GA, Davis SM. The spot sign and tranexamic acid on preventing ICH growth--AUStralasia Trial (STOP-AUST): protocol of a phase II randomized, placebo-controlled, double-blind, multicenter trial. Int J Stroke. 2014 Jun;9(4):519-24. doi: 10.1111/ijs.12132. Epub 2013 Aug 26. PMID 23981692
- [Derived] Pandian JD, Phillips A, Verma SJ, Arora D, Dhasan A, Raju PS, Sylaja PN, Ray BK, Chakraborty U, Johnson J, Sharma PK, Bhoi S, Jha M, Iype T, P C, Khurana D, Ray S, Das D, Kalita N, Adhikari S, Sharma A, Roy J, Sahonta R, Singh S, Chaudhary V, Menon G, Aaron S, Bal D, Dhamija RK, Chaturvedi M, Maheshwari S, Saroja AO, Naik KR, Bhutani N, Dhankhar K, Sharma D, Bhatia R, Gorthi SP, Sarmah B, Pamidimukkala V, Saravanan S, Narayan S, Basumatary LJ, Sundarachary NV, Upputuri AK, Karadan U, Pradeep Kumar VG, Parthasarathy R, Doshi D, Wagh S, Ramakrishnan T, Akhtar S, Desai S, Borah NC, Das R, Mittal G, Jain A, Alapatt PJ, Kulkarni GB, Menon D, Raja P, Puri I, Nambiar V, Yerasu MR, Jaiswal SK, Zirpe K, Gurav S, Sharma S, Kumaravelu S, Benny R, Thakkar V, Pathak A, Kempegowda M, Chander P, Ramrakhiani N, Ks AD, Sarma PS, Huilgol R, Sharma M, Dhaliwal RS. Indian Trial of Tranexamic acid in Spontaneous Intracerebral Hemorrhage study protocol. Int J Stroke. 2025 Jul;20(6):756-762. doi: 10.1177/17474930241307933. Epub 2025 Jan 3. PMID 39633570